CLINICAL TRIAL: NCT04615364
Title: Genetic Evolution of Arboviruses in New Caledonia Between 1995 and 2024 and Impact of Wolbachia
Acronym: DENWOLUTION
Status: Recruiting | Type: Observational
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur de Nouvelle-Calédonie (Unknown); Centre Hospitalier Territorial de Nouvelle-Calédonie (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-022
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Arbovirus Infections; Dengue; Zika; Chikungunya
Keywords: New Caledonia
MeSH Terms: conditions — Arbovirus Infections; Dengue; Zika Virus Infection; Chikungunya Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Arboviruses, diseases transmitted to humans by the bite of an insect vector, are a major public health problem, especially in tropical and sub-tropical countries. A promising strategy aimed at blocking the circulation of arboviruses is to release Aedes aegypti mosquitoes carrying the endosymbiotic bacterium Wolbachia. In 2019, the Wolbachia strategy was implemented in Nouméa as part of the World Mosquito Program. This intervention will modify the epidemiological profile of arboviruses in New Caledonia.

Epidemiological surveillance of arboviruses requires molecular characterization of the virus contained in the serum obtained from the blood collected from patients. This molecular characterization by RNA isolation techniques, RT-qPCR monitoring and sequencing allows the construction of phylogenetic trees.

In the context of the implementation of the World Mosquito Program in Nouméa, the investigators plan to follow the molecular evolution of arboviruses, over the period preceding the releases of mosquitoes carrying Wolbachia (from 1995 to 2019) then over a period of 5 years. following the releases.

At the same time, the virus can be isolated by cell culture techniques and in vitro infections, allowing its study in vitro in cells or in vivo in mosquitoes. This study allows us to measure the impact of the Wolbachia strategy on the evolution of the virus's ability to replicate in cells in the presence of Wolbachia and to be transmitted by the mosquito.

DETAILED DESCRIPTION:
Collection of blood samples from patients with arbovirus infection

This study is a non-interventional study with retrospective part.

This study will improve :

* the assessment of the molecular evolution of arboviruses in the period preceding the implementation of the Wolbachia strategy
* the knowledge of the impact of Wolbachia on the diversity and molecular evolution of arboviruses
* the understanding of arbovirus transmission and replication mechanisms in the presence of Wolbachia

ELIGIBILITY:
Inclusion Criteria:

* Appearance of clinical signs suggestive of an infection with an arbovirus in the 7 days preceding the blood sample,
* Diagnostic confirmation by RT-qPCR of mono-infection with dengue virus or another arbovirus.
* Patients or their representative (s) informed of the possible secondary use for research purposes of the samples initially taken for diagnostic purposes and their derivatives, and who have not since expressed their opposition to the secondary use of the samples diagnostics or their derivatives for research,

Exclusion Criteria:

* Documented opposition from a patient or his representative (s)
* Previously established viral load too low.
* Sample obtained from a sample taken more than 7 days after the appearance of clinical signs of infection.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient infected by arboviruses
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2025-07-17 (Estimated); Study Completion 2025-07-17 (Estimated)

PRIMARY OUTCOMES:
arbovirus genome sequencing | 5 years
  Whole genome sequencing of virus extracted of blood samples from patients collected from 1995 to 2024
genetic evolution of arbovirus strains | 5 years
  bioinformatical analysis of the genome of the strains of arbovirus contained in serum samples collected from 1995 to 2024

SECONDARY OUTCOMES:
measurement of the impact of Wolbachia on the virus genetic evolution | 5 years
  comparison of viral genomes extracted from blood samples collected from 1995 to 2024
measurement of the ability of these viruses to replicate in the presence of Wolbachia | 5 years
  infection of cell lines with virus strains isolated and amplified from patient blood samples collected from 1995 to 2024

CONTACTS AND LOCATIONS:
Overall Officials: Myrielle Dupont-Rouzeyrol, PhD, Principal Investigator — Institut Pasteur de Nouvelle-Calédonie
Locations (1):
- Centre Hospitalier Territorial, Dumbéa Sur Mer, Nouvelle-Calédonie, France

REFERENCES:
- [Derived] Inizan C, Minier M, Prot M, O'Connor O, Forfait C, Laumond S, Marois I, Biron A, Gourinat AC, Goujart MA, Descloux E, Sakuntabhai A, Tarantola A, Simon-Loriere E, Dupont-Rouzeyrol M. Viral evolution sustains a dengue outbreak of enhanced severity. Emerg Microbes Infect. 2021 Dec;10(1):536-544. doi: 10.1080/22221751.2021.1899057. PMID 33686914